CLINICAL TRIAL: NCT00323518
Title: A Phase II Randomized Double Blind Placebo Controlled Trial to Assess Safety and Efficacy of Velafermin for Prevention of Oral Mucositis in Hematologic Cancer Patients Receiving Autologous Stem Cell Transplant
Brief Title: A Phase II Controlled Trial of Velafermin for Prevention of Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CuraGen Corporation (Industry)
Responsible Party: Sponsor
Organization: Celldex Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CG53135-CLN-12
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Oral Mucositis; Stomatitis
Keywords: oral mucositis; hematologic; autologous stem cell transplant; velafermin; stomatitis; oncology - supportive care; mouth diseases
MeSH Terms: conditions — Stomatitis; Mouth Diseases | interventions — FGF20 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): placebo
  Interventions: Drug: placebo
- 2 (Experimental): 30 mcg/kg velafermin
  Interventions: Drug: velafermin
- 3 (Experimental): 10 mcg/kg velafermin
  Interventions: Drug: velafermin
- 4 (Experimental): 60 mcg/kg velafermin
  Interventions: Drug: velafermin

INTERVENTIONS:
Drug: velafermin — administered intravenously as 100mL single dose over 15 minutes on day 1
  Other Names: CG53135-05
  Arms: 2; 3; 4
Drug: placebo — administered intravenously as 100mL single dose over 15 minutes on day 1
  Arms: 1

SUMMARY:
CG53135-05 (velafermin), a recombinant human fibroblast growth factor-20 (rhFGF-20) protein, is under investigation for the prevention of oral mucositis. Oral mucositis is a commonly occurring side effect of high-dose chemotherapy in patients undergoing autologous hematopoietic stem cell transplant. The objective of this Phase II trial is to confirm the safety and efficacy of CG53135-05 (velafermin) when administered as a single dose to patients at risk for developing oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients with multiple myeloma or lymphoma receiving myeloablative CT with or without TBI that require autologous stem cell support. The CT regimens are limited to high dose melphalan (200 mg/m2) as a single agent, BEAM, or TBI with cyclophosphamide or VP-16.
* Adequate organ function that meets institutional requirements for autologous stem cell transplant. A minimum CD34+ cell dose of 2X106 /kg based on ideal body weight (IBW) has been or will be infused.
* ECOG Performance Score of 2 or less
* Signed Informed Consent Form (ICF)

Exclusion Criteria:

* Premenopausal female patients who are pregnant, lactating or are likely to become pregnant
* Patients diagnosed with active sero-positive acquired immunodeficiency syndrome (AIDS) or Hepatitis B/ C
* Patients with known hypersensitivity to recombinant protein therapeutics
* Patients who have taken velafermin (CG53135-05) previously
* Patients who have taken palifermin in the past 90 days
* Patients who have taken other investigational drugs in the past 30 days
* Patients who have untreated symptomatic dental infection
* Patients with a history of sensitivity or allergy to E. coli-derived products
* Patients with WHO Grade 3 or 4 OM at the time of randomization
* Patients who are sensitive or allergic to G-CSF, Fluconazole or acyclovir or equivalent
* Patients with altered mental status precluding understanding of the informed consent process and/or completion of the necessary assessments
* Patients with baseline creatinine level greater than or equal to 3 or any patient with renal insufficiency requiring dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
the incidence of grade 3/4 oral mucositis using WHO grading system | evaluated throughout the study

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Comprehensive Cancer Center, Berkley, California
  - Research Facility, La Jolla, California
  - Scripps Green Medical Center, La Jolla, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Louisiana State University Health Science Center, Shreveport, Louisiana
  - Wayne State University, Detroit, Michigan
  - MAYO Clinic, Rochester, Minnesota
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cornell Medical Center, New York, New York
  - Biomedical Research Alliance of New York, New York, New York
  - Biomedical Research Alliance of New York, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Legacy Good Samaritan Hospital and Cancer Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase-Temple Bone Marrow Transplant Program, Philadelphia, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Medical College of Wisonsin, Milwaukee, Wisconsin